CLINICAL TRIAL: NCT03217357
Title: Effects of Transcranial Direct Current Stimulation on Stress Reactivity and Decision Making in Unaffected Siblings of Patients With Schizophrenia
Brief Title: tDCS, Stress and Risk for Schizophrenia
Acronym: 3S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2017-A00850-53
Record Dates: First submitted 2017-07-05; First posted 2017-07-14 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia
Keywords: tDCS, non invasive brain stimulation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: In a randomized controlled double blind study, 30 subjects, first-degree relatives of schizophrenic patients, were randomly assigned to 2 groups. A group of 15 participants will receive 30 minutes of active tDCS (2mA, 30 minutes with the anode at the left DLPFC and the cathode at the right DLPFC); A group of 15 participants will receive 30 minutes of placebo stimulation. During this stimulation session, all participants will undergo a standardized stress test combining psychosocial stress and physical stress
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject will be blind of the treatment he receives (active or placebo).
  - The experimenter will also be blinded from stimulation (active or placebo) Each subject will be assigned a randomization code, corresponding to the code to enter the tDCS device. This system allows the person who administers tDCS and the subject receiving the stimulation to be blind .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial stimulation in direct current(tDCS)active (Active Comparator): 30 minutes of active Transcranial stimulation in direct current
  Interventions: Device: Transcranial stimulation in direct current
- Transcranial stimulation in direct current(tDCS) placebo (Placebo Comparator): 30 minutes of placebo stimulation
  Interventions: Device: Transcranial stimulation in direct current

INTERVENTIONS:
Device: Transcranial stimulation in direct current — tDCS (2mA, 30 minutes with the anode at the left DLPFC and the cathode at the right DLPFC) active or placebo

SUMMARY:
An exacerbated response to stress mediated by activation of the Hypothalamo-Pituitary-Adrenocortical (HPA) axis is thought to play an important role in the onset, worsening and relapse of schizophrenia. Subjects at risk for schizophrenia (unaffected siblings of patients) displayed an intermediate hyperreactivity to stress as compared with patients and healthy controls.

Symptoms of schizophrenia can be reduced with noninvasive brain stimulation (NIBS) applied over the dorsolateral prefrontal cortex (DLPFC). Importantly, this same DLPFC NIBS protocol can modulate decision making processes and modulate biological reactivity to stress by decreasing salivary cortisol concentration in acute stress condition.

DETAILED DESCRIPTION:
The objective of this project is to evaluate how the modulation of DLPFC activity in acute stress condition influences decision-making in unaffected siblings of patients with schizophrenia.

Methods: 30 unaffected siblings of patients with schizophrenia will be enrolled and randomized into 2 groups. 15 subjects will receive active tDCS (2mA, 30 min, anode left DLPFC, cathode right DLPFC) and 15 will receive sham tDCS.

tDCS procedure: There is a total of 30 minutes of stimulation at the intensity of 2mA (ramp up and ramp down: 30 sec). Sham stimulation consists in delivering 1 minute of real stimulation. The stimulation site (DLPFC) will be anatomically determined according to 10/20 EEG system (F3 & F4). This procedure is in accordance with international guidelines for safety. Safety and blinding will be assessed using specific tools at the end of the protocol.

Stress paradigm: In order to induce moderate stress in humans in laboratory condition, the investigators will use the Maastricht Acute Stress Test (MAST). This test is a combination between physical (hand immersion in cold water) and cognitive (arithmetic calculation) stress. Test will start 5 minutes after the beginning of stimulation session.

Decision-making paradigm: The decision-making task will be performed before and after the MAST (during the stimulation) in order to compare changes induce by stress and/or stimulation. The choose test is the Delay Discounting Task (DDT) permitting a measure of decision-making, reward seeking and impulsivity.

Stress measure: Saliva samples will be collected using a Salivette®, samples will be stored frozen (- 20°C). Saliva cortisol levels will be measured by ELISA. The investigators also will measure heart rate, systolic and diastolic blood pressures at each time of saliva extraction (each 15 minutes, 1st sample at 9:00 am, please see figure 1). Anxiety will be assessed using the State-Trait Anxiety Inventory (STAI) before and after stimulation

ELIGIBILITY:
Inclusion Criteria:

* Subject to genetic risk of schizophrenia, related first-degree schizophrenic patient
* Man and woman
* Age between 18 and 30 years old

Exclusion Criteria:

* Contraindications to the practice of the tDCS, for safety measure, we will use the same contraindications as the practice of the Magnetic resonance imaging
* Psychiatric disorder on axis I of DSM 5
* Pregnant or nursing women

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Cortisol | One year
  Salivary cortisol will be analyzed, using Salivette tubes

SECONDARY OUTCOMES:
Decision-making capacities | 6 mois
  Decision-making capacities will be measured using a computerized version of the delay discounting task in which participants have to choose between 2 rewards
electroencephalography | 6 mois
  EEG will be acquired twice. It consists in an at rest recording of EEG 64 channels, eyes closed to measure spectral power intensities

CONTACTS AND LOCATIONS:
Overall Officials: D AMATO THIERRY, MD - PhD, Principal Investigator — CH LE VINATIER
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No